CLINICAL TRIAL: NCT03500380
Title: A Randomized, Controlled, Multi-center Phase II Clinical Study to Evaluate the Efficacy and Safety of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate for Injection in the Treatment of HER2-positive Locally Advanced or Metastatic Breast Cancer and Phase III Clinical Study to Evaluate the Efficacy and Safety of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate for Injection in the Treatment of HER2-positive Advanced Breast With Liver Metastases
Brief Title: A Study of RC48-ADC Administered Intravenously to Patients With HER2-Positive Metastatic Breast Cancer With or Without Liver Metastases
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C006
Record Dates: First submitted 2018-04-08; First posted 2018-04-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasms; Breast Diseases; Capecitabine; HER2-positive Breast Cancer; HER2 Positive Breast Carcinoma; HER2-positive Advanced Breast With Liver Metastases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RC48-ADC (Experimental): Participants will receive RC48-ADC 2.0 mg/kg intravenous (IV) infusion each 14-day treatment cycle until disease progression (PD) (as assessed by the investigator), unmanageable toxicity, or study termination.
  Interventions: Drug: RC48-ADC
- Lapatinib + Capecitabine (Active Comparator): Participants will receive lapatinib 1250 mg orally once daily during each 21-day cycle + capecitabine 2000 mg/m^2 orally daily on Days 1-14 of each 21-day treatment cycle until PD (as assessed by the investigator), unmanageable toxicity, or study termination.
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: RC48-ADC — RC48-ADC 2.0 mg/kg IV every 14 days
  Other Names: RC48
  Arms: RC48-ADC
Drug: Lapatinib — Lapatinib 1250 mg orally once daily during each 21-day cycle.
  Arms: Lapatinib + Capecitabine
Drug: Capecitabine — Capecitabine 2000 mg/m^2 orally daily on Days 1-14 of each 21-day treatment cycle.
  Arms: Lapatinib + Capecitabine

SUMMARY:
This is a randomized, open, parallel-controlled, multicenter, phase II/III, seamless design clinical trial to compare the efficacy and safety of RC48-ADC with capecitabine + lapatinib in locally advanced or metastatic human epidermal growth factor receptor 2 (HER2) positive breast cancer and HER2-positive advanced breast cancer with liver metastasis.

ELIGIBILITY:
Inclusion criteria for the first phase randomized control period:

* Voluntarily agree to participate in the study and sign the informed consent form.
* Subjects aged 18 - 70 years (inclusive), and the subject who have not reached the age of 71 years old will be considered to be ≤ 70 years of age.
* Expected survival ≥ 12 weeks.
* ECOG PS score 0 or 1.
* Female subjects should be surgically sterilized or in post-menopausal status, or agree to use at least one medically accepted contraceptive methods (such as intrauterine device, contraceptive drug or condom) during study treatment period and for up to 6 months after the study treatment is completed, and the blood pregnancy test must be negative within 7 days prior to study enrollment, and they must not be lactating. For male subjects: all the subjects should be surgically sterilized or agree to use one of the medically approved contraceptive methods during the study treatment period and for an additional of 6 months after the end of the study treatment period.
* Able to understand study requirements, willing and able to comply with study protocol and follow-up procedures.

With Adequate Organ Function

* Bone marrow function:

Hemoglobin ≥ 9 g/dL; Absolute neutrophil count ≥ 1.5×109/L; Platelets ≥ 100 × 109/L;

* Liver function (based on the normal values specified by study site):

Serum total bilirubin ≤ 1.5 × the upper limit of normal (ULN); Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 2.5 × ULN in the absence of liver metastases, while ALT, AST and ALP ≤ 5 × ULN in the presence of liver metastases;

* Renal function (based on the normal values specified by study site):

Serum creatinine ≤ 1.5 × ULN, or creatinine clearance (CrCl) ≥ 60 mL/min as calculated by Cockcroft-Gault formula, or 24-hour urine Crcl ≥ 60 mL/min;

* Cardiac function:

New York Heart Association (NYHA) classification < Grade III; Left ventricular ejection fraction ≥ 50%; Tumor Related Criteria

* Histologically and/or cytologically confirmed invasive locally advanced or metastatic breast cancer that is incurable and unresectable;
* Positive HER2 expression (positive defined as: IHC 3+ or FISH+); previous test results of HER2 expression provided by the subjects (have to be confirmed by the investigator) and those obtained from the study site or the central laboratory were both acceptable; subject are able to provide samples from primary or metastatic tumor sites for HER2 test (either paraffin blocks, paraffin-embedded sections, or sections prepared using freshly excised tissues);
* With prior taxane therapy (monotherapy or in combination with other drugs, treatment duration should be ≥ 2 cycles);
* With prior adjuvant therapy, have received treatment with trastuzumab or its biosimilar for patients with locally advanced cancer or metastasis during relapse and metastasis (monotherapy or in combination with other drugs, such as for ≥ 3 months in the adjuvant therapy phase, and ≥ 6 weeks in the post-relapse and metastatic phase);
* With evidence of tumor progression during or after the most recent treatment as confirmed by the investigator or with documented history;
* No more than 2 lines of chemotherapy received after relapse/metastasis. The number of chemotherapy lines is restricted to chemotherapeutic drugs, and each chemotherapy regimen is counted as a number of chemotherapy line, excluding targeted drugs and/or endocrine drugs; the same maintenance treatment as the previous chemotherapy regimen will not be counted.
* With at least one measurable lesion per RECIST v1.1.

Exclusion Criteria for Randomized Controlled Period in Stage I:

* Use of investigational drugs within 4 weeks prior to study treatment;
* Have received major surgeries within 4 weeks prior to study treatment and have not recovered yet;
* Have received a live vaccine inoculation within 4 weeks prior to the start of study drug administration or was scheduled to receive any vaccine during the study;
* Have experienced arterial/venous thromboembolic events, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism within 1 year prior to the initiation of study treatment;
* Suffering uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, cirrhosis, etc.;
* Currently suffering from active infections requiring systemic treatment;
* With history of active tuberculosis;
* With positive HIV test result;
* Patients with active hepatitis B or C (HBsAg positive and HBV DNA positive; HCVAb positive);
* Presence of effusion in the third space (including massive hydrothorax or ascites) that cannot be controlled by drainage or other methods;
* With known hypersensitivity or delayed-type hypersensitivity to certain components of RC48-ADC, capecitabine, lapatinib or similar drugs;
* With pre-existing gastrointestinal disorders that may affect absorption, such as ileus, ulcerative colitis, chronic diarrhea, inability to swallow, and other conditions that may affect drug administration and absorption;
* With known psychiatric disorders or drug abuse disorders that might have an impact on compliance with protocol requirements;
* Have any other diseases, metabolic disorders, abnormal physical examination findings or abnormal laboratory test results, which, judged by the investigator, are reasonably to suspect a disease or condition as a contraindication of the study drug, or may interfere the interpretation of the study results in the future, or that put the patient at a high risk;
* Women who are pregnant or during lactation period or women/men with childbearing plans;
* Subjects who are estimated to have poor compliance with the clinical study or the investigator determines that there are other factors not appropriate to participate in the study;
* Presence of brain metastases and/or carcinomatous meningitis.
* Had any other malignancy within 5 years prior to signing of the informed consent (except for non-melanoma skin cancer, cervix carcinoma in situ or other tumor that have been effectively treated and considered to be cured);
* Have received prior chemotherapy, radiotherapy, immunotherapy within 4 weeks prior to the first dose of the study drug;
* Have received hormonal therapy for breast cancer within 2 weeks prior to the start of study treatment;
* Patients who received palliative radiotherapy for bone metastases within 2 weeks before the start of study treatment;
* Have received anti-tumor traditional Chinese medicine within 2 weeks prior to the start of study treatment;
* Have received capecitabine within 6 months prior to the start of study treatment, or have failed to respond to prior treatment with capecitabine (including progression while on capecitabine treatment or maintenance of clinical efficacy for a period of less than 6 months after treatment), or with intolerance to capecitabine. Patients who have received capecitabine as adjuvant therapy and have discontinued this therapy for ≥ 6 months are eligible;
* The toxicity of prior anti-tumor therapy had not recovered to CTCAE [Version 4.03] Grade 0-1, with the following exceptions: a). alopecia; b). pigmentation; c). long-term toxicity caused by radiotherapy, which are considered as irreversible by the investigator;
* With prior systemic therapy with or participation in clinical studies with HER2 tyrosine kinase inhibitors (TKIs);
* With prior treatment with T-DM1 or had participated in clinical studies with same class of drugs.
* With known hypersensitivity to 5-fluorouracil or known dihydropyrimidine dehydrogenase deficiency.

Inclusion Criteria for Stage 1 Cross-over Period：

* Had previously participated in the study of randomized controlled period and received lapatinib plus capecitabine, and received no anti-tumor treatment after disease progression (RECIST v1.1 criteria);
* The general situation part refers to the selection criteria of the first stage randomized control period.

Exclusion Criteria for Cross-over Period in Stage I：

* Have received major surgeries within 4 weeks prior to study treatment and have not recovered yet;
* Have received a live vaccine inoculation within 4 weeks prior to the start of study drug administration or was scheduled to receive any vaccine during the study (except the COVID-19 vaccine);
* Have experienced arterial/venous thromboembolic events, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism within 1 year prior to the initiation of study treatment;
* Suffering uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, cirrhosis, etc.;
* Currently suffering from active infections requiring systemic treatment;
* With positive HIV test result;
* Patients with active hepatitis B or C (HBsAg positive and HBV DNA positive; HCVAb positive);
* Presence of effusiona in the third space (including massive hydrothorax or ascites) that cannot be controlled by drainage or other means;
* With known hypersensitivity or delayed-type hypersensitivity to certain components of RC48-ADC or similar drugs;
* With known psychiatric disorders or drug abuse disorders that might have an impact on compliance with protocol requirements;
* Have any other diseases, metabolic disorders, abnormal physical examination findings or abnormal laboratory test results, which, judged by the investigator, are reasonably to suspect a disease or condition as a contraindication of the study drug, or may interfere the interpretation of the study results in the future, or that put the patient at a high risk;
* Women who are pregnant or in lactation period or women/men with childbearing plans;
* Subjects who are estimated to have poor compliance with the protocol of this cross-over period or the investigator determines that there are other factors not appropriate to participate in the study;
* Presence of brain metastases and/or carcinomatous meningitis. Have received prior treatment for brain metastases may be considered for participating in this study, provided that the diseases were stable, had no disease progression as confirmed by imaging examinations within 4 weeks prior to the first dose of the investigational product (IP), and that all neurological symptoms have recovered to baseline level without any evidence of newly emerging or spread brain metastases; moreover, treatment with radiation, surgery or steroids was discontinued at least 14 days prior to the first dose of study drug. This exception did not include cancerous meningitis, which should be excluded regardless of the stability of its clinical status;
* Patients who received palliative radiotherapy for bone metastases within 2 weeks before the start of study treatment;
* Received treatment with lapatinib and/or capecitabine within 2 weeks prior to the first dose of the study drug;
* The toxicity of prior anti-tumor therapy had not recovered to CTCAE [Version 4.03] Grade 0-1, with the following exceptions: a). alopecia; b). pigmentation; c). long-term toxicity caused by radiotherapy, which are considered as irreversible by the investigator;

Inclusion Criteria for Randomized Controlled Period in Stage II：

* The general situation part refers to the selection criteria of the first stage randomized control period.

Exclusion Criteria for Randomized Controlled Period in Stage II：

* The toxicity of prior anti-tumor therapy had not recovered to CTCAE [Version 5.0] Grade 0-1, with the following exceptions: a). alopecia; b). pigmentation; c). long-term toxicity caused by radiotherapy, which are considered as irreversible by the investigator;
* The remaining parts refer to the exclusion criteria of the first stage randomized control period.

Inclusion Criteria for Cross-over Period in Stage II：

* Had previously participated in the study of randomized controlled period and received lapatinib plus capecitabine, and received no anti-tumor treatment after disease progression (RECIST v1.1 criteria);
* Expected survival ≥ 12 weeks;
* ECOG PS score 0 or 1;
* Female subjects should be surgically sterilized or in post-menopausal status, or agree to use at least one medically accepted contraceptive methods (such as intrauterine device, contraceptive drug or condom) during study treatment period and for up to 6 months after the study treatment is completed, and the blood pregnancy test must be negative within 7 days prior to study enrollment, and they must not be lactating. For male subjects: all the subjects should be surgically sterilized or agree to use one of the medically approved contraceptive methods during the study treatment period and for an additional of 6 months after the end of the study treatment period.
* Able to understand study requirements, willing and able to comply with study protocol and follow-up procedures.

With Adequate Organ Function

* Bone marrow function:

Hemoglobin ≥ 9 g/dL; Absolute neutrophil count ≥ 1.5×109/L; Platelets ≥ 100 × 109/L;

* Liver function (based on the normal values specified by study site):

Serum total bilirubin ≤ 1.5 × the upper limit of normal (ULN); Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 2.5 × ULN in the absence of liver metastases, while ALT, AST and ALP ≤ 5 × ULN in the presence of liver metastases;

* Renal function (based on the normal values specified by study site):

Serum creatinine ≤ 1.5 × ULN, or creatinine clearance (CrCl) ≥ 60 mL/min as calculated by Cockcroft-Gault formula, or 24-hour urine Crcl ≥ 60 mL/min;

* Cardiac function:

New York Heart Association (NYHA) classification < Grade III; Left ventricular ejection fraction ≥ 50%;

Exclusion Criteria for Cross-over Period in Stage II：

* The toxicity of prior anti-tumor therapy had not recovered to CTCAE [Version 5.0] Grade 0-1, with the following exceptions: a. alopecia; b. pigmentation; c. long-term toxicity caused by radiotherapy, which are considered as irreversible by the investigator;
* The remaining parts refer to the exclusion criteria of the first phase of the crossover period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by an IRC | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response was assessed by an IRC according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by Investigator | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Tumor response was assessed by investigator according to RECIST v1.1.
Objective Response Rate （ORR） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR).
Duration of Objective Response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  DOR was defined as the time from first documented OR to first documented PD or death from any cause, whichever occurred earlier.
Clinical Benefit Rate （CBR） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Participants were considered as experienced clinical benefit if they had an OR or maintained stable disease (SD) for at least 6 months from randomization. OR: CR or PR determined on 2 consecutive tumor assessments >/=4 weeks apart.
Time to Treatment Failure | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time to treatment failure was defined as the time from randomization to discontinuation of treatment for any reason, including PD (per investigator review), treatment toxicity, or death from any cause.
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 48 months
  OS was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (67):
- China (67):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - An Yang Cancer Hospital, Anyang
  - Beijing Luhe Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Bin Zhou No.1 People's Hospital, Binzhou
  - Jilin Cancer Hospital, Changchun
  - The First Hospital Jilin University, Changchun
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - The Second Xiyang Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Affiliated Hospital of Chengde Medical University, Chengde
  - West China Hospital,Sichuan University, Chengdu
  - Chongqing University Three gorges Hospital, Chongqing
  - The Southwest Hospital of AMU, Chongqing
  - The Second Hospital of Dalian Medical University, Dalian
  - Fujian Cancer Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-Sen Memorial Hospital, Guangzhou
  - The Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou
  - Guizhou Cancer Hospital, Guiyang
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Ha’erbin
  - Anhui Cancer Hospital, Hefei
  - Anhui Province Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Qilu Hospital of Shandong University, Jinan
  - The First People's Hospital of Jining, Jining
  - Yunnan Cancer Hospital, Kunming
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang
  - Jiangsu Cancer Hospital, Nanjing
  - The Affiliated Tumor Hospital of Guangxi Medical University, Nanning
  - The Second People's Hospital of Neijiang, Neijiang
  - Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Changhai Hospital, Shanghai
  - Shanghai Ruijin Hospital, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Yue Bei People's Hospital, Shaoguan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Bethune Hospital, Taiyuan
  - Shanxi Cancer Hospital, Taiyuan
  - Taizhou Enze Medical Center, Taizhou
  - Tai'an City Central Hospital, Tai’an
  - Tianjin Cancer Hospitial, Tianjin
  - Weihai Municipal Hospital, Weihai
  - Hubei Cancer Hospital, Wuhan
  - Tongji Medical College of HUST, Wuhan
  - Wuhan Union Hospital, Wuhan
  - The First Affiliated Hospital of the Fourth Military University of P.L.A., Xi'an
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xing Tai People's Hospital, Xingtai
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Yanbian University Hospital, Yanbian
  - Yantai Yuhuangding Hospital, Yantai
  - Yuncheng Central Hospital, Yuncheng
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No